CLINICAL TRIAL: NCT03154437
Title: An Open-Label, Multicenter, Expanded Access Program for Emicizumab in Patients With Hemophilia A With Inhibitors
Brief Title: An Expanded Access Program of Emicizumab in Participants With Hemophilia A With Inhibitors
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39356
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Emicizumab — Participants will receive emicizumab at a loading dose of 3 milligrams per kilogram (mg/kg) per week subcutaneously (SC) for 4 weeks, followed by a maintenance dose of 1.5 mg/kg per week SC thereafter. Treatment with emicizumab will continue until unacceptable toxicity, withdrawal of consent, participant or physician decision to discontinue treatment, death, the participant is able to obtain commercial drug after emicizumab becomes commercially available, or the sponsor decides to discontinue emicizumab clinical development, whichever occurs first.
  Other Names: ACE910; CH5534262

SUMMARY:
This open-label, multicenter expanded access program (EAP) is designed to provide emicizumab to eligible participants with hemophilia A with factor VIII (FVIII) inhibitors before it is commercially available in the United States for the indication of hemophilia A with FVIII inhibitors. Discontinuation may occur earlier if participant or physician decides to discontinue treatment or the sponsor discontinues emicizumab clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital hemophilia A of any severity and documented history of high-titer inhibitor (that is [i.e.], greater than or equal to [>/=] 5 Bethesda Units)
* History of treatment with episodic or prophylactic bypassing agents for at least the last 24 weeks
* >/=6 (if on an episodic bypassing agent regimen) or >/=2 (if on a prophylactic bypassing agent regimen) bleeds within 24 weeks prior to screening
* Currently using recombinant activated factor VII (rFVIIa) or are willing to switch to rFVIIa as primary bypassing agent for the treatment of breakthrough bleeds
* Adequate hematologic function, defined as platelet count >/= 100,000 per microliters (mcL) and hemoglobin >/=8 grams per deciliter (g/dL) at screening
* Adequate hepatic and renal function

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than hemophilia A
* Ongoing (or plan to receive during the study) immune tolerance induction (ITI) therapy or prophylaxis with FVIII with the exception of participants who have received a treatment regimen of FVIII prophylaxis with concurrent bypassing agent prophylaxis
* Treatment for thromboembolic disease within 12 months before Day 1 (with the exception of previous catheter-associated thrombosis for which antithrombotic treatment is not currently ongoing) or current signs of thromboembolic disease
* Other conditions (example [e.g.], certain autoimmune diseases) that may increase the risk of bleeding or thrombosis
* High risk for thrombotic microangiopathy (TMA), in the investigator's judgment
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Use of systemic immunomodulators (e.g., interferon or rituximab) at enrollment or planned use during the study, with the exception of antiretroviral therapy
* Treatment with any of the following: An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration before Day 1; A non-hemophilia-related investigational drug within the last 30 days or 5 half-lives before Day 1, whichever is longer; An investigational drug concurrently
* Any serious medical condition, treatment, or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in the study

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (14):
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Rush Medical Center, Chicago, Illinois
  - Tulane Medical Center; Investigational/Research Pharmacy, New Orleans, Louisiana
  - Boston Childrens Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hosp Clinics, Kansas City, Missouri
  - Barnabas Health Newark Beth Israel Medical Center - Pulmonary Hypertension & Lung Transplant Program, Newark, New Jersey
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center - Children's Medical Center Dallas, Dallas, Texas
  - University of Texas Medical School, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Bloodworks Northwest (formerly Puget Sound Blood Center); Hemophilia, Seattle, Washington